CLINICAL TRIAL: NCT05270902
Title: Effect of Haemoadsorption During Cardiopulmonary Bypass on Patients After Heart Transplantation
Brief Title: Haemoadsorption During Heart Transplantation
Acronym: CytoSorbHTX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Martin Bernardi, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1933/2021
Record Dates: First submitted 2022-02-02; First posted 2022-03-08 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Heart Transplantation
Keywords: Heart Transplantation; Cytosorb

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, single-blinded, randomized, controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adsorber Group (Active Comparator): Surgery with CPB will be performed according to institutional standards, depending on indications and surgical preferences.
  For the intervention group (adsorber-group), the CytoSorb adsorber will be installed on the CPB machine in a parallel circuit to the body circulation. The flow through the filter will be driven by a roller pump with 300-400 ml.min-1.
  Interventions: Device: CytoSorb Adsorber
- Control (No Intervention): The control group (no-adsorber group) will be treated similarly, but no filter circuit will be installed.

INTERVENTIONS:
Device: CytoSorb Adsorber — Polymer based adsorber system for the elimination of cytokines
  Arms: Adsorber Group

SUMMARY:
To investigate whether the use of haemoadsorption (HA) on cardiopulmonary bypass during heart transplantation (HTX) has an effect on circulating cytokine levels for the first 120 hours after HTX and induces a decreased inflammatory response, increased anti-inflammatory response or immunosuppressive response. Additionally, the influence of HA on primary graft dysfunction, postoperative cerebral dysfunction, postoperative fluid accumulation, renal dysfunction, duration of mechanical ventilation, length of ICU-stay and 30-day mortality should be investigated

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing heart transplantation

Exclusion Criteria:

* Declined informed consent
* Age < 18 years#
* Receiving antileukocyte drugs
* Receiving TNF-α Blockers, immunosuppressive drugs (e.g. tocilizumab)
* DCD
* Ex-vivo perfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in maximal cytokine peak levels (IL-1β, IL-6, IL-33, TNF-α, IL-10) | 5 days
  Difference in maximal cytokine peak levels in various cytokine levels compared to baseline measured by ELISA

SECONDARY OUTCOMES:
Difference of immunosuppression (TTV) | 30days
  Individual immunosuppression measured by Torque-teno-virus load
Difference of immunosuppression (sST2) | 30days
  Individual immunosuppression measured by sST2 levels
primary graft dysfunction score | 7 days
  Differences in primary graft dysfunction score between both groups
30-day mortality | 30 days
  Differences in 30-day mortality between both groups
Mechanical Ventilation | up to 4 weeks
  Differences in length of mechanical ventilation
Delirium | 5 days
  Differences in Confusion assessment method for the ICU between both groups

CONTACTS AND LOCATIONS:
Overall Officials: Martin H. Bernardi, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Divison of Cardiac Thoracic Vascular Anaesthesia and Intensive Care, Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
after completion of study, the results will be published in a peer reviewed journal